CLINICAL TRIAL: NCT05256095
Title: Thinking in Speech for Children With Autism - Pilot Study
Brief Title: Thinking in Speech for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Barbara Baumann, Research Instructor in Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20060157
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder; Speech
MeSH Terms: conditions — Autism Spectrum Disorder; Speech

STUDY DESIGN:
Intervention Model Description: All participants will receive the Thinking in Speech Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Assignment to Intervention Group (Experimental): This group will begin to receive the intervention immediately upon entering the study. Thinking in Speech is a novel cognitive therapy that helps children with autism independently cope with everyday events that cause stress, by developing their ability to use inner speech. Participants will complete two sessions per week for eight week, for a total of sixteen sessions. Sessions will be conducted by speech-language pathologists who are trained in Thinking in Speech. Sessions will be conducted via a secure Zoom platform.
  Interventions: Behavioral: Thinking in Speech
- Waitlist Assignment to Intervention Group (Experimental): The Waitlist group will begin to receive the intervention 10 weeks after entering the study. Thinking in Speech is a novel cognitive therapy that helps children with autism independently cope with everyday events that cause stress, by developing their ability to use inner speech. Participants will complete two sessions per week for eight week, for a total of sixteen sessions. Sessions will be conducted by speech-language pathologists who are trained in Thinking in Speech. Sessions will be conducted via a secure Zoom platform.
  Interventions: Behavioral: Thinking in Speech

INTERVENTIONS:
Behavioral: Thinking in Speech — Thinking in Speech is a therapy to help children with autism learn to cope with daily stressors and improve their communication.

SUMMARY:
This study examines a cognitive therapy for autistic children, Thinking in Speech. Thinking in Speech helps children with autism independently cope with everyday events that cause stress, by developing their ability to use "inner speech".

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of Thinking in Speech (TiS) in teaching children to identify when they are experiencing a problem and learn to ask for help appropriately.

Participants. Participants will be 20 verbal children, aged 7-11, who have been diagnosed with autism or related neurocognitive disorders. Therapists will be experienced and certified speech-language pathologists (SLPs) who will be trained to use TiS For this grant, investigators will develop a standardized training program that can be administered to community SLPs. Training will consist of background reading and discussions, analysis of past therapy sessions, and practice sessions with individualized feedback provided by a trainer. Training will focus on developing the child's ability to ask for help. Asking for help requires a complex combinations of executive functions and being able to adopt the perspective of another person. Training sessions will be recorded for use in further training development and enhancements. A five-week training program is anticipated.

Procedure: Both training and therapy will be delivered remotely. The therapists will plan to conduct sixteen 30-minute remote therapy sessions over 8 weeks - the actual time frame will depend on the health and scheduling demands of the therapists and children. All TiS sessions will be video-recorded. Children will be randomly assigned to either receive therapy immediately or to be placed on a 10-week wait-list after which they will receive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Verbal language ability as reported by the caregiver
* Ages 7-11
* Prior autism or related neurocognitive diagnosis
* Child proficient in English
* Caregiver proficient in English
* Residing in Pennsylvania
* Access to internet at home

Exclusion Criteria:

* History of major child mental illness (e.g., bipolar, schizophrenia, psychosis)
* Child visual and/or hearing impairment that interferes with his/her ability to participate in therapy

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Emotion Dysregulation Inventory scores to Post-Intervention | Up to 20 weeks
  This measure assesses participants' emotion dysregulation via a 30-item measure. 24 items measure reactivity and 6 items measure dysphoria. A raw score is created by summing the items for each subscale, and ranges from 0-96. Higher scores indicate greater emotion dysregulation and lower scores indicate less emotional dysregulation. Participants will be assessed using this measure at baseline and after therapy is completed.

SECONDARY OUTCOMES:
Number of Thinking in Speech therapy sessions attended among all participants | Up to 20 weeks
  Number of sessions attended will be calculated for each participant
Change from Baseline in Patient-Reported Outcomes Measurement Information System - Anger Measure to Post-Intervention | Up to 20 weeks
  The PROMIS Anger item banks assess self-reported angry mood (irritability, frustration), negative social cognitions (interpersonal sensitivity, envy, disagreeableness), and efforts to control anger. Often associated with episodes of frustration that impede goal-directed behavior, anger is marked by attitudes of hostility and cynicism. Specific components relate to verbal and non-verbal evidence of anger. Physical aggression items are not included. The anger short forms are universal rather than disease-specific. All assess anger over the past seven days. The values are summed to create a total score and scores range from 5-25, with higher scores indicating greater levels of anger and lower scores indicated lower levels of anger.
Change from Baseline in Patient-Reported Outcomes Measurement Information System - Anxiety Short Form to Post-Intervention | Up to 20 weeks
  The PROMIS Anxiety item banks assess self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). Anxiety is best differentiated by symptoms that reflect autonomic arousal and experience of threat. Only one behavioral avoidance item is included in the adult item bank; therefore, behavioral fear avoidance is not fully evaluated. The anxiety measures are universal rather than disease-specific. All assess anxiety over the past seven days. Responses are summed to create a total score ranging from 8-40. Higher scores reflect greater levels of anxiety and lower scores reflect less anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Baumann, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No